CLINICAL TRIAL: NCT02179281
Title: Prevention of Hypoglycaemia With Predictive Insulin Suspend Using Medtronic MiniMed™ 640G Sensor Augmented Insulin Pump in Children - The SportGuard Study
Brief Title: Prevention of Hypoglycaemia With Predictive Insulin Suspend Using Sensor Augmented Insulin Pump in Children
Acronym: SportGuard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SG-01
Record Dates: First submitted 2014-06-28; First posted 2014-07-01 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suspend Before Low feature turned ON (Experimental): MiniMed™ 640G system with the "Suspend Before Low" feature turned ON; continuously set on at 3,6 mmol/L (65 mg/dL). "Suspend On Low" Alert and "Resume Basal Alert" for the SmartGuard group should be set OFF.
  Administered intervention: Medtronic MiniMed™ 640G system
  Interventions: Device: Medtronic MiniMed™ 640G system
- Suspend Before Low feature turned OFF (Active Comparator): MiniMed™ 640G system with the "Suspend Before Low" and "Suspend On Low" features are both turned OFF; "Alert On Low" is set at 65 mg/dL (3,6 mmol/L). "Resume Basal Alert" should be set OFF as well.
  Administered intervention: Medtronic MiniMed™ 640G system
  Interventions: Device: Medtronic MiniMed™ 640G system

INTERVENTIONS:
Device: Medtronic MiniMed™ 640G system — The MiniMed™ 640G system is indicated for the continuous delivery of insulin, for continuous or periodic monitoring of glucose levels in the fluid under the skin, with a feature for a prediction of low or high glucose episodes.

SUMMARY:
The aim of the study is to prove whether the use of the SmartGuard feature of the MiniMed system significantly reduces hypoglycemic excursions and thus provide proactive protection to the user.

DETAILED DESCRIPTION:
This is randomized two-arm parallel controlled open label study that will be conducted at two sites, in Slovenia and Israel. It is an investigator initiated pediatric clinical study.

Study will be conducted on pediatric population during two weeks, following a 3 day Run-in period that will allow the patients to get familiar with study device and CGM (SmartGuard OFF).

Patients will be asked to continuously wear the study device for 14 days, which will be set up by study staff according to randomization in the specific group. They will be provided with a diary for entering their daily activity, food consumption (carb count) and eventual adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by a parent/legal guardian and informed assent signed by the study participant prior study entry
* Diagnosed with Type 1 DM at least 12 months prior to signature of Patient Informed Consent (PIC).
* Age between 8-18 years old (inclusive) at signature of PIC
* Treated by CSII with or without CGM at least 3 months prior to signature of PIC, but no use of LGS for last two weeks prior to signature of PIC.
* HbA1c value at screening visit ≤10%
* Knowledgeable on the use of CSII, administering treatment, adjusting insulin according to diet and exercise
* Performance of an average of four (4) SMBG per day, as evidenced from patient files, or latest insulin pump or glucose meter download
* Treated by the investigator's centre for at least 6 months prior signature of PIC.
* Willing to undergo all study procedures

Exclusion Criteria:

* Hearing or vision impairment so that glucose display and alarms cannot be recognized.
* Alcohol or drug abuse.
* Non-compliance with diabetes self-monitoring and disease management
* Documented cutaneous allergy or disease (allergy to sensor or components of the sensor, psoriasis, staphylococcus, exanthema etc.).
* Any documented concomitant chronic disease known to affect diabetes control (e.g. altered renal function, active cancer undergoing treatment, Crohn's disease, ulcerative colitis, Mb Addison disease) or any concomitant pharmacological treatment that might modify glycemic values (e.g. chronic corticosteroid therapy),
* Eating disorders and morbid obesity (defined as adults: BMI>35 and children BMI > 2 SD for age) as assessed by the investigator.
* Any other medical, social or psychological condition that, in the investigator's opinion, makes the patient unable to comply with the study protocol and all study procedures.
* Patient that does not have a reliable support person.
* Participation in another clinical study, on-going or completed less than 2 months prior to signature of PIC.
* Pregnancy (per investigator judgment, including pregnancy test if necessary)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Significant between-group difference in number of hypoglycemic events | After all patients completed 14 days of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tadej Battelino, PhD, Principal Investigator — University of Ljubljana, Faculty of Medicine
Locations (2):
- Schneider Children's Medical Center of Israel, The Jesse Z and Sara Lea Shafer Institute for Endocrinology and Diabetes, Petah Tikva, Israel
- University of Ljubljana, Faculty of Medicine, Ljubljana, Slovenia

REFERENCES:
- [Derived] Battelino T, Nimri R, Dovc K, Phillip M, Bratina N. Prevention of Hypoglycemia With Predictive Low Glucose Insulin Suspension in Children With Type 1 Diabetes: A Randomized Controlled Trial. Diabetes Care. 2017 Jun;40(6):764-770. doi: 10.2337/dc16-2584. Epub 2017 Mar 28. PMID 28351897